CLINICAL TRIAL: NCT04792580
Title: A Single-Center Randomized Double-Masked Placebo-Controlled Parallel-Group, Study of the Effects and Safety of 5% Lifitegrast Ophthalmic Solution in Subjects With Dry Eye Disease in Ocular Graft-versus-Host Disease
Brief Title: The Effects and Safety of 5% Lifitegrast Ophthalmic Solution in Subjects With Dry Eye Disease in Ocular Graft-versus-Host Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Richard W Yee, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Richard W Yee, MD, Sponsor-Investigator, Yee, Richard W., M.D.
Organization: Yee, Richard W., M.D. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIF606A1US09T
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Graft-versus-host-disease; Ocular Graft-versus-host Disease
Keywords: Ocular surface; Bone marrow transplant; stem cell transplant; ocular Graft-versus-Host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Subjects receive lifitegrast 5% ophthalmic solution twice a day for 4 weeks after a 2 week washout.
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution
- Placebo (Placebo Comparator): Subjects receive the lifitegrast vehicle as placebo twice a day for 4 weeks after a 2 week washout.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — Used twice a day in both eyes for 4 weeks after a 2 week washout.
  Arms: Treatment
Drug: Placebo — Used twice a day in both eyes for 4 weeks after a 2 week washout with the same drops.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical efficacy of 5% lifitegrast ophthalmic solution in subjects with dry eye disease secondary to ocular Graft-versus-Host Disease compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* SANDE questionnaire >40 mm
* Schirmer test without anesthesia >2 mm and <10mm across 5 minutes
* Tear film break-up time (TFBUT) < 10 seconds in the worse eye
* The same eye (eligible eye) must fulfill all the above criteria
* Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units (20/200 Snellen value) in both eyes at the time of study enrollment.
* If a female of childbearing potential, have a negative pregnancy test.
* Only patients who satisfy all Informed Consent requirements may be included in the study. The patient must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients must have been approved by the Institutional Review Board (IRB) / Independent Ethics Committee (IEC) for the current study.
* Patients must have the ability and willingness to comply with study procedures.
* Patients must meet the internationally established criteria for a "probable" or "definite" diagnosis of oGVHD. As an inclusion criterion, a diagnosis of oGVHD is established from the Schirmer's 1 tear test, corneal fluorescein staining, OSDI scores, and conjunctival injection. Severity scores are assigned according to the panels provided by the International Chronic Ocular Graft-versus-Host Disease Consensus Group.
* Ability to speak and understand the English language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments.

Exclusion Criteria:

* Evidence of an active ocular infection, in either eye
* Presence of any other ocular disorder or condition requiring topical medication during the entire duration of study
* History of severe systemic allergy or of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis and/or keratitis other than dry eye
* Intraocular inflammation defined as Tyndall score >0
* Systemic disease (excluding GVHD) not stabilized within 1 month before Screening Visit (e.g. diabetes with glycemia out of range, thyroid malfunction..) or judged by the investigator to be incompatible with the study (e.g. current systemic infections) or with a condition incompatible with the frequent assessment required by the study
* Patient had a serious adverse reaction or significant hypersensitivity to any drug or chemically-related compounds or had a clinically significant allergy to drugs, foods, amide local anesthetics or other materials including commercial artificial tears (in the opinion of the investigator)
* Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

  1. are currently pregnant or,
  2. have a positive result at the urine pregnancy test (Baseline/Day 0) or,
  3. intend to become pregnant during the study treatment period or,
  4. are breast-feeding or,
  5. are not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected - and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or Intra Uterine Device (IUD) - during the entire course of, and 30 days after, the study treatment periods
* Any concurrent medical condition, that in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
* Use of topical cyclosporine, topical corticosteroids or any other topical drug for the treatment of dry eye in either eye within 30 days prior to study enrollment.
* Contact lenses or punctum plug use at any time 30 days prior to or during the study
* History of drug addiction or alcohol abuse
* Any prior ocular surgery (including refractive palpebral and cataract surgery) if within 90 days before the screening visit
* Participation in a trial with a new active substance during the past 6 months
* Participation in another trial study at the same time as the present study.
* Previous use of lifitegrast, 5%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Symptoms questionnaire (SANDE) scores to Week 4 | Baseline to Week 4
  The SANDE score is calculated by taking the square root of the product of the severity of symptoms scores and the frequency of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount or absence of dry eye symptoms.

SECONDARY OUTCOMES:
Change from baseline in Schirmer I test (without anesthesia) to Week 4 | Baseline to Week 4
  Without previously instilling anesthetic drops, the Schirmer strip will be inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding contact with the cornea.
  The patients will be instructed to close their eyes gently. After 5 minutes have elapsed, the Schirmer test strip will be removed and the length of the tear absorption on the strip will be measured (millimeters/5 minutes)

OTHER OUTCOMES:
Change from baseline in Symptoms questionnaire (SANDE) scores for frequency to Week 4 | Baseline to Week 4
  The SANDE score is calculated by taking the square root of the product of the frequency of symptoms score. Each of the two scores ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptom. The endpoint here is the SANDE sub-score for frequency.
Change from baseline in conjunctiva vital staining with lissamine green to Week 4 | Baseline to Week 4
  The Oxford scheme is used for grading the scale of conjunctival damage. Briefly, the observer grades the extent of staining across temporal, nasal and central zones between 0 to 5, with 0 representing no staining and 5 representing severe/maximal staining.
Change from baseline in Tear Film Break-Up Time (TFBUT) to Week 4 | Baseline to Week 4
  TFBUT is measured by determining the time to tear break-up. The TFBUT is performed after instillation of 5 μL of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. The patient is instructed to blink several times to thoroughly mix the fluorescein with the tear film.
  A TFBUT greater than 15 " is considered normal, while a break up time of less than 10" is considered pathological.
Change in OSDI score from baseline to Week 4 | Baseline to Week 4
  The Ocular Surface Disease Index score is a 12-item questionnaire designed to survey the dry eye symptomatology of a given patient. In this case, OSDI will be used to assess whether the study drug affects specific symptoms of dry eye more than others. In other words, OSDI may be used to determine whether patients on the study drug see improvement of gritty sensations, sensitivity to light or burning sensations.
Change in Corneal Staining Score from baseline to Week 4 | Baseline to Week 4
  Corneal staining with fluorescein is measured from 0-3 by the NEI grading scale in any one eye region.

CONTACTS AND LOCATIONS:
Locations (1):
- Richard W Yee, MD PLLC, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: No